CLINICAL TRIAL: NCT06921148
Title: The Utility of Silk Bioprotein as a Wound Dressing in Female-to-Male Double-Incision Mastectomy
Brief Title: Silk Bioprotein as a Wound Dressing for Double-Incision Mastectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Ivan Hadad, Assistant Professor of Clinical Surgery, Indiana University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25905
Record Dates: First submitted 2025-03-28; First posted 2025-04-10 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-04

CONDITIONS: Wound Healing

STUDY DESIGN:
Intervention Model Description: All patients who undergo the intervention will act as their own controls. Patients undergo these surgeries bilaterally, meaning one side of their chest will have the interventional dressing applied, and the other side of their chest will have the control dressing applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sylk Wound Dressing (Experimental): Patients who will be enrolled to this study will act as both the control and experimental group. This is a surgery that is done bilaterally for every patient. On one side of the body, the intervention dressing (Silk bioprotein) will be applied; on the other side of the body, the control dressing (Dermabond/Prineo) will be applied. All patients in the study are both in the control and experimental group given they act as their own controls.
  Interventions: Device: Sylk Wound Dressing
- Dermabond/Prineo Dressing (Experimental): Patients who will be enrolled to this study will act as both the control and experimental group. This is a surgery that is done bilaterally for every patient. On one side of the body, the intervention dressing (Silk bioprotein) will be applied; on the other side of the body, the control dressing (Dermabond/Prineo) will be applied. All patients in the study are both in the control and experimental group given they act as their own controls.
  Interventions: Device: Dermabond/Prineo Dressing

INTERVENTIONS:
Device: Sylk Wound Dressing — Patients will have Silk bioprotein post-surgical dressing on one side of chest wall, and will have Dermabond/Prineo on the other side of chest wall. All patients will act as their own controls for this study. This means that all patients are both in the control group as well as the intervention group, given that these surgeries are bilateral in nature and one side of their chest will receive the interventional dressing and the other will receive the control dressing.
  Arms: Sylk Wound Dressing
Device: Dermabond/Prineo Dressing — Patients will have Silk bioprotein post-surgical dressing on one side of chest wall, and will have Dermabond/Prineo on the other side of chest wall. All patients will act as their own controls for this study. This means that all patients are both in the control group as well as the intervention group, given that these surgeries are bilateral in nature and one side of their chest will receive the interventional dressing and the other will receive the control dressing.
  Arms: Dermabond/Prineo Dressing

SUMMARY:
This study will investigate the utility of Silk bioprotein, an FDA-approved and readily available post-surgical dressing, as a wound dressing for patients undergoing double-incision mastectomy for female-to-male gender affirmation surgery.

DETAILED DESCRIPTION:
Medical adhesive-related skin injuries (MARSIs) affect approximately 1.5 million patients annually in the United States are one of the most overlooked complications of surgery. MARSI is a condition secondary to the use of surgical tapes, dressings, and tissue adhesives which can lead to a host of postoperative complications such as allergic contact dermatitis (ACD), wound dehiscence, surgical-site infections (SSIs), and in extreme cases sepsis. A commonly utilized surgical dressing is the Dermabond and Dermabond/Prineo system. Allergic dermatitis to these dressings is an increasingly reported adverse reaction in multiple surgical specialties; moreover, the FDA has found that approximately 75% of the adverse events reported with Dermabond/Prineo were related to ACD. These dressings are reported to produce mechanical skin tears and blisters, which can damage epidermal cells and compromise the protective skin layer, making patients susceptible to infection and other wound-related complications.

Silk bioprotein dressings have shown promise due to their biocompatibility and regenerative properties, potentially reducing MARSI compared to the Dermabond/Prineo system, which remains a standard choice for many surgical procedures. A plethora of preclinical and clinical studies have demonstrated the safety and efficacy of silk in tissue engineering, and recently only two studies have utilized this technology as a surgical site dressing demonstrating its safety and utility compared to other standard wound dressings such as Dermabond/Prineo. Despite these findings, these recent studies utilized a small cohort of patients and had a relatively diverse patient population in regard to type of surgery performed. Therefore, the comparative efficacy of Silk bioprotein dressing remains undetermined. Silk bioprotein dressings and Dermabond/Prineo are both currently used in the IU Health system as surgical wound dressings.

Double-incision mastectomy, a common procedure for female-to-male gender affirmation surgery, is a relatively standardized procedure in terms of wound dimensions, tissue dissection, and closure tension; additionally, all patients undergoing this procedure by definition will receive bilateral procedures. This uniformity allows for a unique study design where patients can serve as their own internal controls. Prior to the introduction of Silk bioprotein dressings to the IU Health/Eskenazi hospital systems, the majority of these surgical wounds were dressed with Dermabond/Prineo, whereas now it is mixed based on product availability. Our study aims to better elucidate the wound healing outcomes of Silk dressing using a patient population that are not only undergoing a fairly standardized surgical procedure, but could also serve as their own internal controls. Our decision would dress one incision with silk dressings, and the other with Dermabond/Prineo. This approach minimizes variability and imposes minimal risk, ensuring a robust comparison of outcomes between the two dressings, and will add data to the current literature on the utility of silk bioprotein dressings in surgical wound care.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 undergoing double-incision bilateral mastectomy for female-to-male gender affirming surgery with the principal investigator.
* Physicians will be plastic surgeons in the IU Health system

Exclusion Criteria:

* Patients with a history of breast cancer.
* Patients with prior history of breast surgery.
* Patients with a prior history of radiation to the chest wall/breast.
* Patients with medical comorbidities that predispose to poor wound healing (diabetes, nutritional deficiency, smoking, inflammatory disease, chronic steroid use, immune deficiency, morbid obesity).
* Patients with a history of documented allergic reaction to Dermabond/Prineo or Silk Bioprotein dressing, or any of the constituents that make up these dressings.
* Significant acute or chronic medical, neurologic, or illness in the patient that, in the judgment of the Principal Investigator, could compromise subject safety, limit the ability to complete the study, and/or compromise the objectives of the study.
* Physicians not in the IU Health system will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-14 (Estimated)

PRIMARY OUTCOMES:
Medical Adhesive-Related Skin Injury (MARSI) | 12 weeks postoperatively
  This outcome will assess the incidence and time point postoperatively of MARSIs in both dressing types (Silk and Dermabond/Prineo) used on the chest walls of patients enrolled in this study. This will be determined via physical examination and photo documentation of patient surgical incisions.
Timeing of premature removal of postoperative dressing | 12 weeks postoperatively
  This objective will the post-operative time at which dressings are removed due to adverse events and/or intrinsic properties of the dressing falling off prior to what was instructed by the operating surgeon. This will be determined by physical exam or via patient-reported outcomes
Postoperative wound infection and dehiscence | Any time up until 12 weeks postoperatively
  This objective will assess the incidence and time postoperatively of wound dehiscence or infection on the postoperative incisions of patients. This will be determined by clinical examination and documented photographs of patient's incisions.

SECONDARY OUTCOMES:
Subjective wound healing outcome by patient | Patients will have their subjective opinions evaluated 1, 2, 4, and 8-12 weeks post-operatively via phone survey
  Patients will have their subjective impression of how their scars heal via phone survey
Subjective wound healing outcome of scar by blinded plastic surgeons | 12 weeks postoperative
  Plastic surgeons not involved in the study/direct patient care will receive blinded postoperative photos of patient surgical scars to determine which side of chest, if any, had better wound healing/scar outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Hadad, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Health, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers due to concerns regarding patient confidentiality and institutional data use agreements